CLINICAL TRIAL: NCT00889616
Title: Phase 1 Study of the Safety and Immunogenicity of BSAM-2/Alhydrogel +CPG 7909, an Asexual Blood Stage Vaccine for Plasmodium Falciparum Malaria in Adults in the US and in Bancoumana, Mali
Brief Title: Phase I Study of the Safety and Immunogenicity of BSAM-2/Alhydrogel +CPG 7909, an Asexual Blood Stage Vaccine for Plasmodium Falciparum Malaria in Adults in the US and Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 999909134; 09-I-N134
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-07-18

CONDITIONS: Malaria
Keywords: Malaria; Asexual Blood Stafe; Plasmodium Falciparum; Immunogenicity; Safety; Vaccine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Aluminum Hydroxide; ProMune

INTERVENTIONS:
Drug: BSAM2/Alhydrogel + CPG 7909

SUMMARY:
Background:

* Globally, the Plasmodium falciparum parasite is responsible for at least 247 million acute cases of malaria each year, resulting in about 1 million deaths. Approximately 90 percent of these deaths, the majority in children under 5 years of age, occur in Africa due to infection with P. falciparum.
* People living in endemic areas develop natural immunity to P. falciparum as a result of repeated infection. Consequently, children who survive to 5 years of age rarely succumb to life-threatening disease despite frequent infection. This acquired immunity is mediated in part by blood-stage parasite-specific antibodies. Thus, parasite proteins expressed during the blood-stage have been proposed as good candidates for inclusion in a vaccine.
* A number of P. falciparum merozoite antigens have been identified as promising blood-stage vaccine candidates, including Merozoite Surface Protein 1 (MSP 1) and Apical Membrane Antigen 1 (AMA 1). This Phase I study is the first time that the combination vaccine (BSAM-2/Alhydrogel +CPG 7909) will be given to humans. The vaccine will be administered in a randomized, open-label (U.S.)/single-blinded (Mali), dose-escalating trial.

Objectives:

* To assess safety and reactogenicity of the combination vaccine (BSAM-2/Alhydrogel +CPG 7909) in malaria-naive U.S. adults and semi-immune Malian adults.
* To determine the antibody response of the combination vaccine to the AMA 1 and MSP 142 proteins, as measured by antibody levels and parasite growth inhibition.
* To determine the extent to which the antibody response to the individual antigens (AMA 1 and MSP 142) is correlated when the combination vaccine is given, and to determine T and B cell responses to vaccination.

Eligibility:

* United States: Healthy volunteers between 18 and 50 years, inclusive. Available for the 52 weeks of the trial and willing to participate in the study as evidenced by signing the informed consent document.
* Mali: Healthy volunteers between 18 and 45 years, inclusive, and a known resident of the village of Bancoumana. Available for the 52 weeks of the trial; willing to participate in the study as evidenced by signing the informed consent document or by fingerprinting the consent document with the signature of a witness.
* Potential participants must meet extensive health and screening requirements to participate in this study. Good general health is required as a result of review of medical history and clinical testing at the time of screening.
* Women who are pregnant or breastfeeding are not eligible.

Design:

* During the 52-week study, participants will receive the first vaccine and complete the following:

  * Physical examination and patient education regarding the signs and symptoms of potential adverse effects.
  * Blood and urine testing, and vital signs (blood pressure, temperature, heart rate, and respiratory rate).
  * United States: Education on the use of digital thermometer, injection-site reaction measurement, and malaria vaccine side-effect memory enhancement tool (daily symptom diaries).
  * Mali: Additional blood draws for malaria smear and urine test for chloroquine testing.
* U.S. and Mali participants will return to the study site on specified days throughout the 52 weeks to receive two additional vaccines, record vital signs, complete additional blood and urine testing, and review patient education.
* U.S. participants will record oral temperature once during the day, as well as pain, tenderness, redness, swelling at the injection site and any systemic signs or symptoms for 6 days following each immunization.
* Participants will receive financial compensation (United States) or food (Mali) to compensate for their time.

DETAILED DESCRIPTION:
This Phase I study will evaluate the blood stage P. falciparummalaria vaccine candidate BSAM-2/Alhydrogel +CPG 7909 in adults in the US and Mali. BSAM-2 contains a mixture of two proteins found on the surface of merozoites, AMA1 and MSP1(42). The study is open label, dose escalating in the US, and will be single-blinded and randomized with a comparator vaccine (Euvax B - Hepatitis B) in Mali. All volunteers will receive three doses of vaccine, given at 0, 2, and 6 months and administered in the deltoid muscle. The US arm of the study will be conducted at the Center for Immunization Research (CIR), in Washington DC. Fifteen (15) healthy volunteers will receive 40 (micro)g BSAM-2/Alhydrogel +500 (micro)g CPG 7909 at CIR, followed by another 15 who will receive 160 (micro)g BSAM-2/Altlhydrogel +500 (micro)g CPG 7909. Safety data to at least one week after the second vaccination from all US volunteers will be reviewed by a Safety Monitoring Committee prior to vaccinating volunteers in Mali. The highest safe dose will be administered in Mali after safety data in US adults have been reviewed by the SMC. The Mali arm of the study will be conducted in Bancoumana. Thirty (30) volunteers will be randomized to receive either BSAM 2/Alhydrogel +CPG7909 or the licensed comparator vaccine. The primary objective of the study is to demonstrate safety and reactogenicity of the vaccine in both malaria naive and semi-immune adults. Secondary objectives are to determine the antibody response of the combination vaccine to the AMA1 and MSPl(42) proteins, as measured by antibody levels and parasite growth inhibition. Study endpoints are the incidence of local and systemic adverse events, antibody responses to AMA1 and MSP1(42) proteins, and in vitro growth inhibition of falciparum parasites. Exploratory immunologic analyses will also be conducted.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a volunteer to participate in this trial:

* Age between 18 and 50 years (US) or 18 and 45 years (Mali), inclusive
* Good general health as a result of review of medical history and/or clinical testing at the time of screening
* Available for the duration of the trial (52 weeks in the U.S. and 104 weeks in Mali)
* Willingness to participate in the study as evidenced by signing the informed consent document, or by fingerprinting the consent document with the signature of a witness (Mali)
* Known resident of the village of Bancoumana (Mali)

EXCLUSION CRITERIA (US):

A volunteer will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Pregnancy as determined by a positive urine or serum test at any point during the study for human choriogonadotropin (Beta-hCG) (if female).
2. Subject is unwilling to use reliable contraception methods for the period of at least 2 months prior to first vaccination to 3 months after last vaccination (if female). Reliable methods of birth control include: pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; surgical sterilization; vaginal ring; intrauterine device; abstinence; and post-menopause (if female).
3. Currently is lactating and breast-feeding (if female).
4. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol.
5. Neutropenia as defined by an absolute neutrophil count less than 1500/mm(3).
6. Alanine transaminase (ALT) level above the laboratory-defined upper limit of normal.
7. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
8. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the subject unable to comply with the protocol.
9. History of receiving any investigational product within the past 30 days.
10. Participant has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
11. History of a severe allergic reaction or anaphylaxis.
12. Severe asthma. This will be defined as:

    * Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past 2 years, or that requires the use of oral or parenteral corticosteroids
    * Clinically significant reactive airway disease that does not respond to bronchodilators
13. Positive ELISA and confirmatory Western blot tests for HIV-1.
14. Positive ELISA and confirmatory tests for hepatitis C virus (HCV).
15. Positive hepatitis B surface antigen (HBsAg) by ELISA.
16. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren s syndrome, or autoimmune thrombocytopenia.
17. Known immunodeficiency syndrome.
18. Positive serum anti-dsDNA titer.
19. Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
20. Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
21. History of a surgical splenectomy.
22. Receipt of blood products within the past 6 months.
23. Previous receipt of an investigational malaria vaccine.
24. Receipt of antimalarial prophylaxis during the past 12 months, or receipt of chloroquine or related compounds (hydroxychloroquine, amodiaquine, or primaquine) in the 8 weeks prior to study entry.
25. Prior malaria infection by history.
26. Any medical, psychiatric, social, or occupational condition or other responsibility that, in the judgment of the Principal Investigator (PI), would interfere with the evaluation of study objectives.

EXCLUSION CRITERIA (MALI):

A volunteer will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Pregnancy as determined by a positive urine (Beta-hCG test at any point during the study (if female).
2. If female, subject and her spouse have not used or are unwilling to use reliable contraceptive methods such as: abstinence, birth control pills or birth control patches or vaginal ring, diaphragm with spermicide, IUD (intrauterine device), condom with spermicide, progestin implant or injection, or surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation) prior to enrollment to 3 months after the final vaccination. (At the time of vaccination, a female subject must have had a negative urine pregnancy test on 2 occasions at least 2 weeks apart, and must have used a reliable contraceptive method in the interim.)
3. Currently is lactating and breast-feeding (if female).
4. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, chronic infectious or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
5. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
6. Pre-existing known autoimmune diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren s syndrome, autoimmune thrombocytopenia.
7. Laboratory evidence of possible autoimmune disease determined by anti-dsDNA titer that equals or exceeds 25 IU.
8. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25 times the upper limit of normal of the testing laboratory).
9. Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing confirmed by repeat testing of clean-catch, midstream sample). (More than trace blood on urine dipstick will not exclude a female who is actively menstruating.)
10. Laboratory evidence of hematologic disease (absolute leukocyte count less than 3000/mm(3) or greater than 11,500/mm(3); hemoglobin less than 0.9 times the lower limit of normal of the testing laboratory, by gender; absolute granulocyte count less than 1300/mm(3); absolute lymphocyte count less than 1000/mm(3); or platelet count less than 110,000/mm(3).
11. Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
12. Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.
13. Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
14. History of a severe allergic reaction or anaphylaxis.
15. Severe asthma. This will be defined as:

    * Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past 2 years, or that requires the use of oral or parenteral corticosteroids
    * Clinically significant reactive airway disease that does not respond to bronchodilators
16. Positive hepatitis B surface antigen (HBsAg). Hepatitis C antibody by rapid diagnostic test.
17. Known immunodeficiency syndrome.
18. Use of systemic corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
19. Receipt of a live vaccine within past 4 weeks or a non-live vaccine within past 2 weeks prior to entry into the study.
20. History of a surgical splenectomy.
21. Receipt of blood products within the past 6 months.
22. Previous receipt of an investigational malaria vaccine.
23. History of use of chloroquine or related compounds (hydroxychloroquine, amodiaquine, or primaquine) within 8 weeks of study entry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2009-04-23; Study Completion 2012-07-18 (Actual)

PRIMARY OUTCOMES:
To assess safety and reactogenicity of BSAM-2/Alhydrogel + CPG 7909 in malaria-naive US adults and semi-immune Malian adults.

SECONDARY OUTCOMES:
To determine the antibody response of the combination vaccine to the AMA1-1 and MSP1(42) proteins, as measured by antibody levels and growth inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth D Ellis, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Johns Hopkins University, Baltimore, Maryland, United States
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Sachs J, Malaney P. The economic and social burden of malaria. Nature. 2002 Feb 7;415(6872):680-5. doi: 10.1038/415680a. PMID 11832956
- [Background] Richie TL, Saul A. Progress and challenges for malaria vaccines. Nature. 2002 Feb 7;415(6872):694-701. doi: 10.1038/415694a. PMID 11832958
- [Background] Healer J, Crawford S, Ralph S, McFadden G, Cowman AF. Independent translocation of two micronemal proteins in developing Plasmodium falciparum merozoites. Infect Immun. 2002 Oct;70(10):5751-8. doi: 10.1128/IAI.70.10.5751-5758.2002. PMID 12228305
- [Derived] Ellis RD, Wu Y, Martin LB, Shaffer D, Miura K, Aebig J, Orcutt A, Rausch K, Zhu D, Mogensen A, Fay MP, Narum DL, Long C, Miller L, Durbin AP. Phase 1 study in malaria naive adults of BSAM2/Alhydrogel(R)+CPG 7909, a blood stage vaccine against P. falciparum malaria. PLoS One. 2012;7(10):e46094. doi: 10.1371/journal.pone.0046094. Epub 2012 Oct 4. PMID 23056238